CLINICAL TRIAL: NCT06412367
Title: FUNCTIONAL ASSESSMENT FOR SURGERY BY A TIMED WALK
Acronym: FAST Walk
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Duminda Wijeysundera, MD PhD FRCPC FAHA, Unity Health Toronto
Other Study IDs: 23-065
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Surgery-Complications; Postoperative Complications
Keywords: Six Minute Walk Test; Functional assessment
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The FAST Walk study aims to determine whether a walking test called the 6-minute walk test (6MWT) can help identify people who are more likely to experience complications after surgery. This test will be completed before surgery. We hope that the results of this study will help improve care for patients having major surgery in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years
2. ≥1 risk factors for postoperative complications
3. Elective non-cardiac surgery with expected post-surgery stay ≥2 days
4. Preoperative 6MWT is feasible
5. Working knowledge of official language(s) in country of study recruitment

Exclusion Criteria:

1. Endovascular surgery
2. Lower limb orthopedic surgery
3. Contraindications to 6MWT

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample will include adults who warrant preoperative risk assessment for inpatient non-cardiac surgery. To identify patients at elevated risk for complications, participants must be aged ≥40 y and have ≥1 risk factor for postoperative complications.
Sampling Method: Non-Probability Sample
Enrollment: 1672 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after surgery
  Major postoperative complications grade II to V in Clavien-Dindo scheme

SECONDARY OUTCOMES:
Days alive and out of the hospital | 30 days after surgery
  Postoperative functional recovery measured counting number of days patient is alive and not in hospital
Significant new disability | 90 days after surgery
  Postoperative functional recovery measured by new disability after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Duminda N Wijeysundera, MD PhD FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wijeysundera DN, Salbach NM, Chan MTV, Alibhai SMH, Puts MTE, Jerath A, Khadaroo R, Ehtesham S, Pazmino-Canizares J, Ladha KS, Granton JT, Amado L, Duceppe E, Hladkowicz E, Lee SM, Macdonell SY, Parotto M, Perlas A, Serrano PE, Thorleifson MD, van Vlymen JM, van Waes J, Racz E, Wilmhurst L, McIsaac DI; FAST Walk Study Investigators. Functional Assessment for Surgery by a Timed Walk (FAST Walk) study: protocol for a multicentre prospective cohort study of the 6 min walk test for preoperative risk stratification in major non-cardiac surgery. BMJ Open. 2026 Jan 5;16(1):e113111. doi: 10.1136/bmjopen-2025-113111. PMID 41490857